CLINICAL TRIAL: NCT02117336
Title: A Phase I/Ib Study of P1446A-05 in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL).
Brief Title: Clinical Study of Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision not related to patient safety
Sponsor: Piramal Enterprises Limited (Industry)
Collaborators: Dana-Farber Cancer Institute (Other); Norris Cotton Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1446A-05/79/13
Record Dates: First submitted 2014-04-08; First posted 2014-04-17 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P1446A-05 (Experimental)
  Interventions: Drug: P1446A-05

INTERVENTIONS:
Drug: P1446A-05 — The study have dose escalation phase, followed by a dose extension phase.
  * Dose escalation phase: five Dose Levels will be evaluated in the 'dose escalation' phase. The Dose Levels selected are 50 mg (Dose Level 1), 75 mg (Dose Level 2), 125 mg (Dose Level 3), 200 mg (Dose Level 4) and 275 mg (Dose Level 5), once daily. If required, a 25 mg once daily dose (Dose Level -1) will also be studied. For Dose Levels 1, 2 and 3 there will be 2- dosing periods: Single Dose and Continuous Dose. At least 3-patients will be enrolled at each Dose Level. Dosing regimens planned for Dose Level 4 and 5 are 200 and 275 mg once daily. In the continuous dose period, patients will receive P1446A-05 on a 28-day cycle, until the occurrence of disease progression or unacceptable toxicity.
  * Dose Extension Phase: Up to a total of 14 patients will be treated at the MTD of P1446A-05, determined in the dose escalation phase, until the occurrence of disease progression or unacceptable toxicity or death.

SUMMARY:
This is an open-label, Phase I/Ib trial with a dose escalation phase, followed by a dose extension phase. The objective of the dose escalation phase is to evaluate the pharmacokinetics (PK) and MTD of P1446A-05 in relapsed/refractory CLL and the objective of the dose extension phase is to evaluate the safety, efficacy and pharmacodynamics of P1446A-05 in 14 patients at the MTD level.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or flow cytometry confirmed diagnosis of B-cell chronic lymphocytic leukemia/small lymphocytic lymphoma (B-CLL/SLL) according to the IWCLL 2008 criteria. The malignant B cells must co-express CD5 with CD19 or CD20. Patients who lack CD23 expression on their leukemia cells should be examined for (and found NOT to have) either t(11;14) or cyclin D1 overexpression, to rule out mantle cell lymphoma.
2. Active disease meeting at least 1 of the following IWCLL 2008 criteria for requiring treatment:

   * A minimum of any one of the following constitutional symptoms:

   Unintentional weight loss >10% within the previous 6 months prior to screening Extreme fatigue (unable to work or perform usual activities) Fevers of greater than 100.5ᵒF for ≥2 weeks without evidence of infection Night sweats without evidence of infection.
   * Evidence of progressive marrow failure as manifested by the development of, or worsening of anemia or thrombocytopenia
   * Massive (i.e., >6 cm below the left costal margin), progressive or symptomatic splenomegaly
   * Massive nodes or clusters (i.e., >10 cm in longest diameter) or progressive lymphadenopathy
   * Progressive lymphocytosis with an increase of >50% over a 2-month period, or an anticipated doubling time of less than 6 months
   * Autoimmune anemia or thrombocytopenia that is poorly responsive to corticosteroids
3. Patients with relapsed/refractory CLL defined as having received ≥2 treatment regimens that included:

   * A treatment regimen containing cytotoxic agents (eg, fludarabine, pentostatin, cladribine, cyclophosphamide, chlorambucil, bendamustine) AND
   * A treatment regimen containing a therapeutic anti-CD20 antibody (e.g., rituximab, ofatumumab, obinutuzumab) AND
   * A treatment regimen containing ibrutinib unless patient is not a candidate
   * All treatment regimens must have been administered for ≥2 cycles unless patient is immediately allergic or intolerant to the regimen
   * A disease expert at the study site must have a detailed discussion with the patient of other treatment options which either have been approved by the FDA or are part of or relevant to the standard care of patients with B-CLL/SLL in the multiply relapsed setting
4. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0-2
5. Patients ≥18 year old
6. Patients must have organ function as defined below:

   * Direct bilirubin ≤2 X institutional ULN (unless due to known Gilbert's syndrome or compensated hemolysis directly attributable to CLL)
   * AST or ALT less than or equal to 2.5 X institutional ULN
   * Creatinine ≤1.5 mg/dL OR estimated creatinine clearance ≥60 mL/min calculated using Cockcroft-Gault equation
   * Total white blood cell count ≤200,000/mm3
   * Platelets ≥10,000/mm3 with no active bleeding
7. Ability to understand and the willingness to sign a written informed consent document
8. Ability to swallow and retain oral medication
9. Patients receiving chronic or acute warfarin treatment are not excluded, but should be monitored very closely or considered for switch to other therapies. P1446A-05 is both highly protein bound and a competitive inhibitor of CYP2C9 at higher concentrations and thus may potentiate the action of warfarin in patients
10. Women of childbearing potential must have a negative serum β-human chorionic gonadotropin or urine pregnancy test at screening
11. All patients of reproductive potential (heterosexually active men and women) must agree to a use of a barrier method of contraception and a second method of contraception and men must agree not to donate sperm during the study and for at least 4 weeks after receiving the last dose of study treatment

Exclusion Criteria:

1. Recent therapeutic intervention including a) prior nitrosoureas or mitomycin C; prior radio- or toxin-immunoconjugates within 6 weeks; b) therapeutic anticancer antibodies (including rituximab, ofatumumab and obinituzumab) within 4 weeks; and c) all other chemotherapy or radiation therapy within 2 weeks prior to initiation of study drug
2. The patient has not recovered from adverse events related to prior therapy to Grade ≤1 (excluding Grade 2 alopecia and neuropathy)
3. Chronic use of corticosteroids in excess of prednisone 20 mg/day or its equivalent
4. Patients who have been in the past enrolled on a study of a Cdk inhibitor
5. History of prior malignancy except: a) Malignancy treated with curative intent and no known active disease present for ≥2 years prior to initiation of current study; b) adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; c) adequately treated in situ carcinomas (e.g., cervical, esophageal, breast, etc.) without evidence of disease; d) asymptomatic prostate cancer managed with "watch and wait" strategy; e) myelodysplastic syndrome which is clinically well controlled and no evidence of the cytogenetic abnormalities characteristic of myelodysplasia on the bone marrow at screening
6. Patients with uncontrolled immune hemolysis or thrombocytopenia (positive direct antiglobulin test in absence of hemolysis is not an exclusion)
7. Patients with known Richter's transformation which is progressive and is deemed to require immediate chemotherapy (history of Richter's transformation is not an exclusion); patients with prolymphocytic leukemia (prolymphocytes in blood >55%)
8. Patients with clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic conditions which manifest with diarrhea, refractory nausea, vomiting or any other condition that will interfere significantly with the absorption of study drugs
9. Patients with mean QTc interval >450 msec at screening and patients taking drugs known to prolong the QTc interval (see Section 9, Appendix D) who cannot be switched to an alternative drug
10. Nursing woman
11. Known history of Human Immunodeficiency Virus (HIV) or active Hepatitis B or C. Intravenous immunoglobulin (IVIG) can cause a false positive hepatitis B serology. If patients receiving routine IVIG have core antibody or surface antigen positivity without evidence of active viremia (negative hepatitis B DNA) they may still participate in the study, but should have hepatitis serologies and Hepatitis B DNA monitored periodically by the treating physician.
12. Any condition for which participation in the study is judged by the Investigator to be detrimental to the patient with inter-current illness including, but not limited to an uncontrolled active infection; unstable angina pectoris; uncontrolled cardiac arrhythmia; transient ischemic attack or pulmonary embolism during the previous 1 month or psychiatric/social situations that would jeopardize compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Cycle 1 (Day 1 to 28 )
  * To establish maximum tolerated dose (MTD) of P1446A 05 in patients with relapsed/refractory chronic lymphocytic leukemia (CLL).
  * There will be two phase, a dose escalation phase, followed by a dose extension phase.
  * In the 'dose extension phase', up to a total of 14 patients will be treated at the MTD of P1446A-05, determined in the 'dose escalation' phase, until the occurrence of disease progression or unacceptable toxicity or death
Dose Limiting Toxicity | Cycle 1 (Day 1 to 28 )
  To establish dose limiting toxicities (DLTs) of P1446A 05 in patients with relapsed/refractory chronic lymphocytic leukemia (CLL).
  - There will be two phase, a dose escalation phase, followed by a dose extension phase.

SECONDARY OUTCOMES:
Overall response | At the end of every 2 cycles,Until disease progression or unacceptable toxicity (average of 2years)
  * To determine the efficacy (overall response ) of P1446A 05 in patients with relapsed/refractory CLL.
  * Overall Response will be assessed according to IWCLL 2008 criteria.
  * Kaplan-Meier curve of overall survival will also be presented. OS will be evaluated in the dose extension phase only.
Progression-free survival | At the end of every 2 cycles, until disease progression or unacceptable toxicity (average of 2years)
  * To determine the efficacy (progression-free survival) of P1446A 05 in patients with relapsed/refractory CLL.
  * Kaplan-Meier estimates of progression-free survival i.e. median and inter-quartile range will be presented.
  * Kaplan-Meier curve of overall survival will also be presented. OS will be evaluated in the dose extension phase only.
Pharmacokinetic profile (Cmax,Tmax and AUC) | SD1, Cycle1-Cycle 5 (average of 5 month)
  * Samples for pharmacokinetic analysis for PK profile (Cmax,Tmax and AUC) will be collected on S-D1at pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 h post on Day S-D1 of single dose period (for Dose Levels 1, 2 and 3).
  * In the continuous dose period, samples will be collected on Day 28 of Cycle 1 at pre-dose, and at 0.5, 2, 4, 6, 8 and 24 h post-dose. Additional samples will be collected pre dose on Day 15 and 22 of Cycle 1 to monitor the attainment of steady state. Pre-dose samples will also be collected on C2D15, C2D28, C3D15, C3D28 and C5D1.
  * PK parameters will be obtained using standard non-compartmental methods.
  * PK evaluations will not be performed in the dose extension phase.
  * Descriptive statistics will be provided for the PK parameters. The PK analysis will be performed using WinNonlin software

OTHER OUTCOMES:
Biomarker Analysis | Cycle1Day1, Cycle1Day28, Until disease progression or unacceptable toxicity (average of 2years)
  To assess whether established (IGHV, p53 and Notch mutational status and ZAP70 and CD38 expression,) and exploratory biomarkers (e.g. expression levels of Cyclin D1, p53 etc.) predict response to P1446A-05 in relapsed/refractory CLL

CONTACTS AND LOCATIONS:
Overall Officials: Dr Alexey V Danilov, MD, PhD, Principal Investigator — Dartmouth-Hitchcock Norris Cotton Cancer Centre; Dr Jennifer R Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock Norris Cotton Cancer Centre, Lebanon, New Hampshire